CLINICAL TRIAL: NCT03295656
Title: Contrast-Enhanced Ultrasound Diagnosis of Acute Appendicitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unanticipated delays.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Harriet Joan Paltiel, Associate Professor of Radiology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00025591
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IV Contrast-Enhanced US (Experimental): IV sulfur hexafluoride lipid-type A microspheres, 0.03 mL/kg, 2 doses per examination, total dose not to exceed 4.8 mL. Single examination per patient.
  Interventions: Drug: Sulfur hexafluoride lipid-type A microspheres

INTERVENTIONS:
Drug: Sulfur hexafluoride lipid-type A microspheres — Contrast-enhanced US imaging of the appendix
  Other Names: Lumason

SUMMARY:
This study evaluates the ability of contrast-enhanced ultrasound to improve the diagnosis of acute appendicitis in children compared to conventional ultrasound.

DETAILED DESCRIPTION:
Acute appendicitis is the most common surgical emergency in children. Diagnostic evaluation for possible appendicitis frequently leads to imaging studies. Magnetic resonance imaging (MRI) and computed tomography (CT) are currently the gold-standard techniques for the diagnosis or exclusion of acute appendicitis. However, these methods not always immediately available; may require administration of intravenous contrast material with the potential for allergic reactions and nephrotoxicity; and, in the case of CT, requires the administration of ionizing radiation that is linked to the long-term development of radiation-induced cancers. The current study will evaluate a potentially safer, radiation-free diagnostic method for acute appendicitis, using contrast-enhanced ultrasound to provide a more accurate means of visualizing the appendix than conventional US imaging.

ELIGIBILITY:
Inclusion Criteria:

* Children who have had a conventional abdominal US study to rule out acute appendicitis and are scheduled for an MRI or CT examination.

Exclusion Criteria:

* Children with serious comorbid conditions, including but not restricted to severe cardiac, pulmonary, renal, or hepatic disease; prior bone marrow or solid organ transplant; cancer; or presence of a ventriculoperitoneal shunt.
* Children with an allergy to either the active or inactive components of Lumason.
* Pregnant or nursing patients.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Contrast-enhanced ultrasound diagnosis of acute appendicitis | One week
  The efficacy of contrast-enhanced US in improving the diagnosis of acute appendicitis compared to conventional US will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Paltiel, MDCM, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No